CLINICAL TRIAL: NCT02089386
Title: Tamoxifen to Treat Barrett's Metaplasia
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201404013
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Barrett Metaplasia
MeSH Terms: conditions — Barrett Esophagus | interventions — Tamoxifen; Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tamoxifen (Experimental): Tamoxifen 20 mg daily for 12 weeks
  Interventions: Drug: Tamoxifen; Procedure: Endoscopy

INTERVENTIONS:
Drug: Tamoxifen
  Other Names: Nolvadex®; Soltamox®
Procedure: Endoscopy

SUMMARY:
Treat Barrett's esophagus (BE) patients with tamoxifen to Barrett's metaplasia as measured by changes in Barrett's esophagus appearance by endoscopy and histology as well as changes in SOX2 and CDX2.

DETAILED DESCRIPTION:
Treat Barrett's esophagus (BE) patients with tamoxifen to determine the effects on Barrett's metaplasia as measured by changes in Barrett's esophagus appearance by endoscopy and histology. Tamoxifen treatment may induce SOX2 expression, decrease CDX2 and promote esophageal stem cell activity, leading to regression of Barrett's metaplasia. To test this hypothesis, we will conduct a prospective, pilot study where patients with BE, without high grade dysplasia, are treated with tamoxifen and assessed for changes in the appearance of their BE by endoscopy and histology as well as changes in the SOX2/CDX2 ratio indicative of an improvement in BE metaplasia

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven Barrett's esophagus that is non-dysplastic or with low grade dysplasia.
* At least 18 years of age.
* ECOG performance status ≤ 2
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥1,500/mcl
  * Platelets ≥ 100,000/mcl
  * AST(SGOT)/ALT(SGPT) ≤1.5 x IULN
  * Serum creatinine within normal institutional limits or less than the lower limit of normal institutional limits; or creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Prior history of esophageal cancer.
* Prior history or current use of tamoxifen or anti-estrogen therapy.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to tamoxifen.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. Female patients must have a negative urine pregnancy test within 14 days of study entry.
* Known HIV-positivity and on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with tamoxifen. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Taking medications known to affect drug metabolism via the CYP3A4, CYP2C9, or CYP2D6 pathways.
* History of blood clots (i.e. pulmonary embolism, DVTs).
* Concurrent use of anticoagulants (i.e. Coumadin/warfarin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-07-09 (Actual); Primary Completion 2016-06-21 (Actual); Study Completion 2016-06-21 (Actual)

PRIMARY OUTCOMES:
Extent of Barrett's involvement and changes in histology | End of 12 weeks (at the time of second endoscopy)
  The biopsy procedures with 4 quadrant biopsies/2 cm for histology and additional biopsies for freezing for macromolecular analysis to assess the preliminary diagnostic value of this marker pair in identifying levels of metaplasia in BE and as an indicator of response to tamoxifen treatment. The tissue from the two endoscopic procedures will be assessed for changes in the following related to tamoxifen therapy.

SECONDARY OUTCOMES:
Changes in SOX2 and CDX2 expression | End of 12 weeks (at the time of second endoscopy)
  The main outcome measurements are SOX2 and CDX2, analyzed as a ratio. We will use a one sample paired non-parametric Wilcoxon test to test the significant difference if the ratio difference is not normally distributed. Normality assumption can be examined by visual Q-Q plot and formal Kolmogorov-Smirnov statistic. In addition, we will explore the patient level characteristics on treatment effect using a linear regression model. Specifically, we will use the difference ratio as the response variable and patient characteristics of interest as explanatory variables. Regression coefficients associated with the explanatory variables quantify the effect of these variables on the difference ratio, with t or F statistic testing for the statistical significance.
Tolerance of tamoxifen | 4 months (30 days after cessation of tamoxifen or after second endoscopy - whichever occurs later)
  As measured by toxicities using CTCAE version 4.0
Changes in the length of Barrett's esophagus involvement | End of 12 weeks (at the time of second endoscopy)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Mills, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindblad M, Garcia Rodriguez LA, Chandanos E, Lagergren J. Hormone replacement therapy and risks of oesophageal and gastric adenocarcinomas. Br J Cancer. 2006 Jan 16;94(1):136-41. doi: 10.1038/sj.bjc.6602906. PMID 16404367
- [Background] Huh WJ, Khurana SS, Geahlen JH, Kohli K, Waller RA, Mills JC. Tamoxifen induces rapid, reversible atrophy, and metaplasia in mouse stomach. Gastroenterology. 2012 Jan;142(1):21-24.e7. doi: 10.1053/j.gastro.2011.09.050. Epub 2011 Oct 14. PMID 22001866
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu